CLINICAL TRIAL: NCT05952193
Title: Evaluation of the POSOS Device for Iatrogenesis Detection in Clinical History? A Vignettes Study
Acronym: YGenHiVi
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Centre Hospitalier de Bourg en Bresse (Other); Saint Antoine University Hospital (Other); CHU de Rouen - Accueil (Other); CHU de Créteil (Unknown); Médipôle Lyon-Villeurbanne (Other); Centre Hospitalier Universitaire de Nice (Other); University Hospital, Montpellier (Other); University Hospital, Lille (Other); Centre Hospitalier de Niort (Other); Centre Hospitalier Régional Metz-Thionville (Other); University Hospital, Grenoble (Other); CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PI2023_843_0070
Record Dates: First submitted 2023-07-11; First posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-06

CONDITIONS: Iatrogenesis; Clinical Vignettes; Diagnostic Performance Study; Medical Information Search; Artificial Intelligence
Keywords: Iatrogenesis; Clinical vignettes; Diagnostic performance study; Medical Information Search; Artificial Intelligence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- seniority ≥3 years + POSOS
- seniority ≥3 years without POSOS
- seniority <3 years with POSOS
- seniority <3 years without POSOS

SUMMARY:
This study is a multicenter evaluation of diagnostic performance using simulated clinical vignettes. It aims to test the effectiveness of the POSOS app in detecting drug-induced iatrogenesis in urgent medical situations, an issue of public health importance. Participating physicians, who are randomly assigned to either use or not use POSOS, are categorized based on their years of experience. Vignettes, including a mixture of complex, simple, and non-iatrogenesis cases, are assigned to these doctors. During the simulation, physicians respond to their respective vignettes on the YgheniVi platform, with responses recorded at two intervals (5 min and 15 min). The supervising physicians subsequently fill out an e-CRF, providing further data on the time spent, the number of medical research applications used, and the overall user experience of POSOS. A doctor/pharmacist pair then corrects the answers to the vignettes.

ELIGIBILITY:
Inclusion Criteria:

* Not applicable as the study population is made up of clinical vignettes, there is no inclusion of patients.
* The physicians included are emergency physicians, selected by convenience so as to have as many physicians (seniority of practice 3 years after thesis) as (seniority of practice less).

Exclusion Criteria:

* Not applicable.
* Simulations with technical faults will be excluded: (absence of the test doctor, internet access not working, PC malfunction, serious disruptions during the simulation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The physicians included are emergency physicians, selected by convenience so as to have as many physicians (seniority of practice 3 years after thesis) as (seniority of practice less).
Sampling Method: Non-Probability Sample
Enrollment: 128 (Estimated)
Dates: Start 2023-06-21 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
the proportion of overall correct responses in each groups | 5 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No